CLINICAL TRIAL: NCT00868374
Title: Quetiapine XR Monotherapy or Adjunctive Therapy to Antidepressants in the Treatment of Major Depressive Disorder With Comorbid Generalized Anxiety Disorder
Brief Title: Quetiapine Extended Release (XR) Treatment of Major Depressive Disorder With Comorbid Generalized Anxiety Disorder
Acronym: MDD/GAD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to low enrollment
Sponsor: Keming Gao (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Keming Gao, Director, Mood and Anxiety Clinic, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-07-29
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Quetiapine XR
  Interventions: Drug: Quetiapine XR
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine XR — Days 1-14 - 50 mg/day; Days 14-21 - 100mg/day; Day 21-End of Study - 150mg/day
  Other Names: Seroquel
  Arms: 1
Drug: Placebo — Days 1-14 - 50 mg/day; Days 14-21 - 100mg/day; Day 21-End of Study - 150mg/day
  Arms: 2

SUMMARY:
The primary objective is to test the hypothesis that quetiapine XR (Extended Release) monotherapy or adjunctive therapy to antidepressant is superior to placebo monotherapy or placebo adjunctive therapy to antidepressant(s) in the acute treatment of depression symptoms in patients with MDD and comorbid GAD. The secondary objectives are to test the hypotheses that quetiapine XR is superior to placebo in the reduction of anxiety symptoms in patients with major depressive disorder and comorbid generalized anxiety disorder, the improvement of the quality of sleep in patients with major depressive disorder and comorbid generalized anxiety disorder and the improvement of the quality of life in patients with major depressive disorder and comorbid generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent before beginning any study-specific procedures
* Male and female patients at least 18 years of age - 70 years of age
* Meets Diagnostic and Statistical Manual IV (DSM-IV) criteria for MDD, currently depressed
* DSM-IV diagnosis of current GAD
* Women with reproductive potential must have a negative urine pregnancy test

Exclusion Criteria:

* Patients who have had a current episode of depression for less than 4 weeks from enrollment
* Patients who have been treated for their current depressive episode for more than 3 weeks with Quetiapine therapy 50 mg/day
* Patients currently taking antidepressants known to cause somnolence/sedation such as mirtazapine or unable to wean off current antidepressant if they choose monotherapy
* Patients who meet DSM-IV criteria for substance dependence confirmed by the Substance Use Disorder Module of the Structured Clinical Interview for DSM-IV (SCID), for any substance except for caffeine and nicotine, with substance abuse within last 3 months or substance dependence within last 6 months;
* Concurrent obsessive-compulsive disorder
* Patients with a history of clinically significant cardiac, renal, neurologic, cerebrovascular, metabolic, or pulmonary disease, or other disease or clinical finding that is unstable or that, in the opinion of the investigator, would be negatively effected by trial medication or that would effect trial medication
* A patient with diabetes mellitus (DM) fulfilling one of the following criteria:

  * Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) > 8.5%
  * Admitted to hospital for treatment of DM or DM related illness within the past 12 weeks
  * Not under physician care for DM
  * Physician responsible for patient's DM care has not indicated that the patient's DM is controlled
  * Physician responsible for patient's DM care has not approved the patient's participation in the study
  * Has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks before randomization (for thiazolidinediones (glitazones) this period should not be less than 8 weeks before randomization)
  * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks

Note: If a patient with DM meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study. A patient could be enrolled at a later time if DM is stabilized.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine XR: Quetiapine XR : Days 1-14 - 50 mg/day; Days 14-21 - 100mg/day; Day 21-End of Study - 150mg/day
- Placebo: Placebo : Days 1-14 - 50 mg/day; Days 14-21 - 100mg/day; Day 21-End of Study - 150mg/day
Period: Overall Study
Arm/Group | Quetiapine XR | Placebo
Started | 12 | 11
Completed | 5 | 4
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 48.3 (11.3) | 41.2 (6.1) | 45.1 (7.1)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 4 | 8 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in 17 Item Hamilton Rating Scale for Depression (HAM-D-17)
Description: The Hamilton Rating Scale for Depression (HAM-D-17) is a 17-item clinician-rated measure that queries symptoms of depression, with a possible total score ranging for 0 to 52. A total score of 0-7 indicates no depression, a total score of 8-12 indicates doubtful depression, a total score of 13-17 indicates mild depression, a total score of 18-24 indicates moderate depression and a total score of 25-52 indicates severe depression.
Time Frame: Week 0 - Week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 12 | 11
units on a scale | -0.5 [-22.1 to 21.1] | 3.9 [-1.5 to 9.4]

ADVERSE EVENTS:
Arm/Group | Quetiapine XR | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 11/12 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine XR (N=12) | Placebo (N=11)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine XR (N=12) | Placebo (N=11)
Dry Mouth (General disorders) | 6 (6) | 1 (1)
Fatigue (General disorders) | 5 (5) | 3 (3)
Headache (General disorders) | 3 (3) | 0 (0)
Sedation (General disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Muscle Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eye Twitching (Eye disorders) | 0 (0) | 1 (1)
Gas (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increase Appetite (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes